CLINICAL TRIAL: NCT02445573
Title: A Pilot Randomized Placebo Controlled Trial of Electroacupuncture for Women With Pure Stress Urinary Incontinence
Brief Title: Efficacy of Electroacupuncture (EA) for Women With Pure Stress Urinary Incontinence (SUI)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Responsible Party: Principal Investigator, huanfang xu, doctor, Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2012BAI24B01-021
Record Dates: First submitted 2015-05-13; First posted 2015-05-15 (Estimated); Results first posted 2015-06-15 (Estimated); Last update posted 2015-06-15 (Estimated); Status verified 2015-05

CONDITIONS: Stress Urinary Incontinence
Keywords: stress urinary incontinence; electroacupuncture; efficacy
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- EA group (Active Comparator)
  Interventions: Other: EA
- Sham EA group (Placebo Comparator)
  Interventions: Other: sham EA

INTERVENTIONS:
Other: EA — When acupuncturing, adhesive pads were first pasted on acupoints after sterilization in either group. In EA group, participants were needled at bilateral BL33 at an angle of 30 to 45 degree inward and downward, and at bilateral BL35 slightly toward upside and outside, to a depth of 50 to 60 mm using acupuncture needles of size 0.30×75 mm. Needles were then lifted, thrusted and twirled evenly for 3 times. Paired electrodes of EA apparatus were attached transversely to bilateral BL33 and BL35 (using real electrodes) respectively, with a continuous wave of 50 Hz and a current intensity of 1-5 milliampere (mA) for 30 min. Participants were treated with EA 3 sessions a week on alternate days for 6 successive weeks.
  Arms: EA group
Other: sham EA — When acupuncturing, adhesive pads were first pasted on acupoints after sterilization in either group. In sham EA group, participants were needled at sham BL33 and sham BL35, which were about 20 mm lateral to BL33 and BL35, respectively, with blunt needle tips piercing adhesive pads and not piercing the surface of the skin, using placebo needles of size 0.30×25 mm. Needles were then lifted, thrusted and twirled evenly for 3 times. Paired electrodes of EA apparatus were attached transversely to bilateral sham BL33 and sham BL35 (using sham electrodes) respectively. The parameters of sham EA apparatus and the treatment course were the same as in the EA group.
  Arms: Sham EA group

SUMMARY:
The purpose of this study is to preliminarily assess the efficacy of electroacupuncture (EA) for women with pure stress urinary incontinence (SUI).

DETAILED DESCRIPTION:
This was a pilot randomized, placebo controlled trial to preliminarily assess the efficacy of EA for women with pure SUI. Eligible participants were randomly assigned to EA group or sham EA group in a 1:1 ratio via a central randomization system by acupuncturists. Participants, outcome assessors and statisticians were blinded to treatment allocation. Subject blinding is achieved via the aid of adhesive pads used in both groups, placebo needle with a blunt tip and sham EA electrode lines. Assuming a two-sided alpha of 0.05, power of 90%, and a 20% drop-out, a sample size of 36 would be needed for each group. The investigators expanded the sample size to 80 cases (40 cases per group) to increase the reliability of the study. The investigators performed statistical analysis based on the intention-to-treat principle. All patients accepting randomization were included in the analysis. Missing data were filled in by the last observed value. Student t tests or Mann-Whitney U tests were used for the comparison of continuous variables; chi-square tests, Fisher's exact tests or Kruskal-Wallis H tests were used to compare categorical variables, as appropriate. For measures collected at two time points, paired t-tests or Wilcoxon signed rank tests were used as appropriate. A statistically significant difference was set at P<0.05.

ELIGIBILITY:
Inclusion Criteria:

* Eligible women were 40 to 75 years of age, and met the clinical diagnosis recommendations of SUI by the International Consultation on Urological Diseases:

  * involuntary urine leakage on effort, exertion, sneezing or coughing which stopped when the stress ends;
  * visible involuntary leakage from the urethra synchronous with increased abdominal pressure, or a pad weight gain >1 g in 1-hour pad test;
  * without symptoms of urinary frequency and urgency.

Exclusion Criteria:

* Women were excluded from the study if they met any of the following criteria: *other type of urinary incontinence (UI) (urge, mixed, or overflow UI, etc);

  * symptomatic urinary tract infection;
  * ever received UI or pelvic surgery;
  * a severity of pelvic organ prolapse ≥ degree 2;
  * residual urinary volume >30 ml;
  * maximum flow rate ≤ 20 ml/s;
  * limited in walking, stairs climbing and running;
  * receiving specialized treatment for SUI, or taking medicine affecting bladder function;
  * serious cardiovascular, cerebral, liver, kidney, or psychiatric disease, diabetes, multiple system atrophy, injury of cauda equina, or myeleterosis;
  * being pregnant or breastfeeding;
  * with cardiac pacemaker, metal allergy or severe needle phobia;
  * unlike to give written formed consent.

Ages: 40 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2012-12; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zhishun Liu, doctor, Principal Investigator — Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Locations (1):
- Guang'anmen hospital of China Academy of Chinese Medical Sciences, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Xu H, Liu B, Wu J, Du R, Liu X, Yu J, Liu Z. A Pilot Randomized Placebo Controlled Trial of Electroacupuncture for Women with Pure Stress Urinary Incontinence. PLoS One. 2016 Mar 9;11(3):e0150821. doi: 10.1371/journal.pone.0150821. eCollection 2016. PMID 26960195

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited through posters and specialist's recommendations in Guang'anmen hospital of China Academy of Chinese Medical Sciences, Beijing, China, from December 2012 to June 2014.
Pre-assignment Details: A total of 181 women with UI were invited to participate in the study. 101 women were excluded from the trial before assignment to groups, of whom 87 did not meet inclusion criteria, 10 declined to participate, 4 were afraid of acupuncture. 80 women were eligible and randomly assigned to EA group (n=40) or sham EA group (n=40).
Period: Overall Study
Arm/Group | EA Group | Sham EA Group
Started | 40 | 40
Completed | 39 | 38
Not Completed | 1 | 2
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Population: All randomized population were included in baseline analysis.
Groups:
- EA Group: EA: When acupuncturing, adhesive pads were first pasted on acupoints after sterilization in either group. In EA group, participants were needled at bilateral BL33 at an angle of 30 to 45 degree inward and downward, and at bilateral BL35 slightly toward upside and outside, to a depth of 50 to 60 mm using acupuncture needles of size 0.30×75 mm. Needles were then lifted, thrusted and twirled evenly for 3 times. Paired electrodes of EA apparatus were attached transversely to bilateral BL33 and BL35 (using real electrodes) respectively, with a continuous wave of 50 Hz and a current intensity of 1-5 mA for 30 min. Participants were treated with EA 3 sessions a week on alternate days for 6 successive weeks.
- Total: Total of all reporting groups
Arm/Group | EA Group | Sham EA Group | Total
Number analyzed (Participants) | 40 | 40 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.05 (7.91) | 57.97 (8.42) | 58.60 (8.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 40 | 80
  Male | 0 | 0 | 0
Educational level [Number; unit: participants]
  Preliminary education and below | 2 | 5 | 7
  Secondary education | 30 | 21 | 51
  Tertiary education | 8 | 14 | 22
Childbearing [Number; unit: participants]
  yes | 40 | 38 | 78
  no | 0 | 2 | 2
Number of births [Number; unit: participants]
  0 | 0 | 2 | 2
  1 | 25 | 25 | 50
  2 | 9 | 7 | 16
  ≥3 | 6 | 6 | 12
Initial childbearing age [Mean (Standard Deviation); unit: years] | 24.65 (2.94) | 23.71 (2.84) | 24.19 (2.91)
Number of vaginal delivery [Median (Inter-Quartile Range); unit: vaginal delivery] | 1.00 [1.00 to 2.00] | 1.00 [1.00 to 2.00] | 1.00 [1.00 to 2.00]
Number of cesarean [Number; unit: participants]
  yes | 0 | 0 | 0
  no | 40 | 40 | 80
Menopause [Number; unit: participants]
  yes | 31 | 30 | 61
  no | 9 | 10 | 19
Hysterectomy [Number; unit: participants]
  yes | 3 | 2 | 5
  no | 37 | 38 | 75
BMI [Median (Inter-Quartile Range); unit: kg/m^2] | 23.44 [22.09 to 25.53] | 22.70 [21.47 to 24.28] | 23.13 [21.66 to 24.63]
Duration of disease [Median (Inter-Quartile Range); unit: years] | 5.04 [2.54 to 8.81] | 5.00 [2.37 to 8.07] | 5.00 [2.67 to 8.32]
Ever received SUI treatment [Number; unit: participants]
  yes | 6 | 2 | 8
  no | 34 | 38 | 72
Severity of SUI rated by amount of urine leakage measured by 1-hour pad test [Number; unit: participants]
  Mild (1.1-9.9 g) | 24 | 32 | 56
  Moderate (10-49.9 g) | 16 | 6 | 22
  Severe (≥50 g) | 0 | 2 | 2
Urine leakage measured by 1-hour pad test [Median (Inter-Quartile Range); unit: g] | 5.30 [2.33 to 16.00] | 4.60 [2.30 to 16.70] | 4.90 [2.30 to 16.20]
72-hour incontinence episode frequency (IEF) [Median (Inter-Quartile Range); unit: episodes] — Number of stress urinary incontinence episodes was collected over the last 72 hours (i.e.,in the last three days) of the week for baseline assessment.
  episodes | 4.00 [2.00 to 6.75] | 5.00 [1.25 to 9.00] | 5.00 [2.00 to 9.00]
International Consultation on Incontinence Questionnaire-Short Form (ICIQ-SF) score [Mean (Standard Deviation); unit: units on a scale] — The International Consultation on Incontinence Questionnaire-Short Form (ICIQ-SF) was a brief and robust measure for evaluating the symptoms and impact of urinary incontinence.It was used to assess the influence of urinary incontinence on quality of life during the past 4 weeks retrospectively. It contained three items on frequency, amount of leakage, and overall impact on quality of life, and a fourth, non-scored item for the assessment of type of incontinence. A total score was summed by the scores of the first three items, ranging from 0 to 21. A higher value indicates increased severity.
  units on a scale | 9.08 (4.24) | 8.80 (4.54) | 8.94 (4.37)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline of Urine Leakage Measured by 1-hour Pad Test
Time Frame: Baseline and week 6
Measure: Median (Inter-Quartile Range); unit: g
Arm/Group | EA Group | Sham EA Group
Number analyzed (Participants) | 40 | 40
g | 2.50 [1.80 to 14.60] | 0.05 [-0.28 to 0.50]

2. Secondary Outcome: Change From Baseline of the 72-hour Incontinence Episode Frequency (IEF)
Description: Data of IEF was from 72-hour bladder diary recorded by participants over the last 72 hours of weeks 0 (baseline), weeks 2, 4, 6 (treatment period) and weeks 15-18,and 27-30 (follow-up period).
  The 72-hour IEF of weeks 1-6 equaled the sum of 72h IEF at weeks 2, 4 and 6 divided by 3; The 72-hour IEF of weeks 15-18 equaled the sum of 72h IEF at weeks 15-18 divided by 4; The 72-hour IEF of weeks 27-30 equaled the sum of 72h IEF at weeks 27-30 divided by 4.
Time Frame: Baseline, weeks 1-6, weeks 15-18 and weeks 27-30
Measure: Median (Inter-Quartile Range); unit: episodes
Arm/Group | EA Group | Sham EA Group
Number analyzed (Participants) | 40 | 40
episodes
  week 6 | 2.00 [0.42 to 3.25] | 0.67 [-0.59 to 2.25]
  week 18 | 3.00 [1.06 to 5.00] | 2.00 [0 to 5.19]
  week 30 | 3.25 [1.25 to 5.69] | 1.00 [-0.69 to 2.88]

3. Secondary Outcome: Change From Baseline of the Total ICIQ-SF Scores
Description: The International Consultation on Incontinence Questionnaire-Short Form (ICIQ-SF) was a brief and robust measure for evaluating the symptoms and impact of urinary incontinence.It was used to assess the influence of urinary incontinence on quality of life during the past 4 weeks retrospectively. It contained three items on frequency, amount of leakage, and overall impact on quality of life, and a fourth, non-scored item for the assessment of type of incontinence. A total score was summed by the scores of the first three items, ranging from 0 to 21. A higher value indicates increased severity.
Time Frame: Baseline, and weeks 6, 18 and 30
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | EA Group | Sham EA Group
Number analyzed (Participants) | 40 | 40
units on a scale
  week 6 | 2.68 (3.19) | 0.16 (2.29)
  week 18 | 5.60 (4.19) | 2.13 (4.20)
  week 30 | 5.89 (4.29) | 1.48 (3.39)

4. Secondary Outcome: Patient Self-evaluation of Therapeutic Effect
Description: Participants were asked to rate the extent of help that they received from treatment as no help, little help. moderate help or great help.
  Number of participants reporting different extent of help was collected.
Time Frame: weeks 6, 18 and 30
Measure: Number; unit: participants
Arm/Group | EA Group | Sham EA Group
Number analyzed (Participants) | 40 | 40
participants
  no-week 6 | 0 | 15
  little-week 6 | 7 | 14
  moderate-week 6 | 11 | 4
  great-week 6 | 22 | 7
  no-week 18 | 1 | 15
  little-week 18 | 5 | 8
  moderate-week 18 | 9 | 5
  great-week 18 | 25 | 12
  no-week 30 | 1 | 17
  little-week 30 | 4 | 11
  moderate-week 30 | 8 | 3
  great-week 30 | 27 | 9

5. Other Pre Specified Outcome: Adverse Events
Description: Number of participants who experienced Adverse Events was collected.
Time Frame: weeks 1-30
Measure: Number; unit: participants
Arm/Group | EA Group | Sham EA Group
Number analyzed (Participants) | 40 | 40
participants
  serious adverse events | 0 | 0
  EA related adverse events | 3 | 2

ADVERSE EVENTS:
Time Frame: 30 weeks
Arm/Group | EA Group | Sham EA Group
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 3/40 | 2/40
OTHER ADVERSE EVENTS (reported when occurring in more than 0.06% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EA Group (N=40) | Sham EA Group (N=40)
hematoma (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
persistent pain after EA (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
fatigue (General disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No